CLINICAL TRIAL: NCT06255587
Title: Relationship Between the Sagittal Lumbopelvic Alignment and Balance Control in Adolescents With Mechanical Low Back Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Manal Helmy Koura, Lecturer, Benha University
Other Study IDs: PT.BU.EC.5
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Low Back Pain, Mechanical
MeSH Terms: conditions — Low Back Pain | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Screening — cross sectional

SUMMARY:
To examine the relationships between lumbopelvic sagittal alignment parameters (lumbar lordosis, sacral slope, pelvic tilt, and pelvic incidence) and balance control in adolescents with mechanical low back pain.

DETAILED DESCRIPTION:
To examine the relationships between lumbopelvic sagittal alignment parameters (lumbar lordosis, sacral slope, pelvic tilt, and pelvic incidence) and balance control in adolescents with mechanical low back pain.Patients will be recruited from the secondary schools in Benha city be general invitations, and the study will be conducted at outpatient clinic of faculty of physical therapy, Benha University

ELIGIBILITY:
Inclusion Criteria:

* age between 15 and 18 years, either sex, and symptoms lasting longer than three months, which imply chronicity

Exclusion Criteria:

* Spinal pathologies or surgery, or any other deformities or visual or auditory issues, as well as ongoing physical or medical treatment for LBP

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents with low back pain
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
level of back pain | 10 minutes
  Visual Analogue scale
standardized lateral views radiographs in a neutral standing position for the lumbopelvic region | 15 minutes
  Lumbar lordosis, sacral slope, pelvic tilt, and pelvic incidence
Balance control | 20 minutes
  Biodex Balance system

IPD SHARING:
Plan to Share IPD: Undecided